CLINICAL TRIAL: NCT01450176
Title: Comparing Patient Satisfaction Throughout the Day With PATADAY (OLOPATADINE HYDROCHLORIDE) 0.2% QD or BEPREVE (BEPOTASTINE BESILATE OPHTHALMIC SOLUTION) 1.5% BID
Brief Title: Comparing Patient Satisfaction With Pataday or Bepreve
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McCabe Vision Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MAC-04-11; 3776-001 (Registry Identifier: Sterling IRB)
Record Dates: First submitted 2011-10-07; First posted 2011-10-12 (Estimated); Last update posted 2014-01-09 (Estimated); Status verified 2014-01

CONDITIONS: Eye Allergies
Keywords: eye; itching; allergies
MeSH Terms: conditions — Pruritus; Hypersensitivity | interventions — Olopatadine Hydrochloride; bepotastine besilate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pataday once daily (Active Comparator): 15 subjects will administer Pataday once daily for 2 weeks. Then these subjects will administer Bepreve twice daily for 2 weeks.
  Interventions: Drug: Olopatadine hydrochloride 0.2%
- Bepreve twice daily (Active Comparator): Bepreve twice daily for 2 weeks, then subjects will use Pataday once daily for 2 weeks
  Interventions: Drug: Bepotastine besilate ophthalmic solution 1.5%

INTERVENTIONS:
Drug: Olopatadine hydrochloride 0.2% — 1 drop in each eye once daily for 2 weeks
  Other Names: Pataday
  Arms: Pataday once daily
Drug: Bepotastine besilate ophthalmic solution 1.5% — 1 drop in each eye twice daily for 2 weeks
  Other Names: Bepreve
  Arms: Bepreve twice daily

SUMMARY:
The purpose of this study is to compare patient satisfaction with Pataday (Olopatadine hydrochloride 0.2%) one daily (QD) and Bepreve (Bepotastine besilate ophthalmic solution 1.5%) two times a day (BID).

DETAILED DESCRIPTION:
5 week randomized study with 15 subjects using Pataday qd for 2 weeks, and the other 15 subjects using Bepreve BID for 2 weeks. Following a one-week washout period, the two groups are given the opposite test article (TA) for 2 weeks. Subjects to complete daily diary regarding effects of drug and are seen in clinic for 3 exams.

ELIGIBILITY:
Inclusion Criteria:

* Be male or female subjects of any racial/ethnic group.
* Be at least 18 years of age or older.
* Have a diagnosis of allergic conjunctivitis with active symptoms, with no concurrent ocular allergy associated conditions and no plans to have ocular surgery during study period.
* Willing and able to return for all required visits and follow instructions from investigator and staff.
* Able to self-administer test article (TA) or have a caregiver available to instill all doses of TA.
* If a woman, capable of becoming pregnant, agrees to have pregnancy testing performed at screening (must be negative) and agrees to use a medically acceptable form of birth control (intrauterine device, birth control pill, patch or subcutaneous implant, condoms, diaphragm, and abstinence) throughout the study duration and for at least one week prior to and one week after completion of the study. Women considered capable of becoming pregnant include all females who have experienced menarche and who have not experienced menopause (as defined by amenorrhea for greater than 12 consecutive months) or have not undergone successful surgical sterilization (hysterectomy, bilateral tubal ligation, or bilateral oophorectomy).
* Sign and date the informed consent form approved by an Institutional Review Board (IRB)/Independent Ethics Committee (IEC).
* Be willing/able to return for all required study visits, to follow instructions from the study investigator and his/her staff, and to complete and return the Screening and Subject Diaries.

Exclusion Criteria:

* Have known hypersensitivity to BEPREVE or PATADAY or any of their components.
* Are actively taking steroids or antihistamines during the study or within 7 days prior to enrolling in the study.
* Are pregnant, planning to become pregnant, or nursing/lactating.
* Have a known history of alcohol or drug abuse.
* Participated in a study of an investigational drug or device within the past 30 days prior to enrolling in the study.
* Have a presence of an active ocular infection (bacterial, viral or fungal), positive history of an ocular herpetic infection, or preauricular lymphadenopathy at any visit.
* Have any significant illness {eg: any autoimmune disease, or severe cardiovascular disease (including arrhythmias)}that the Investigator feels could be expected to interfere with the subject's safety or study parameters and/or put the subject at anyh unnecessary risk.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2011-09; Primary Completion 2011-10 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Relief of ocular itching | 5 weeks
  All day relief of ocular itching throughout the treatment period.

SECONDARY OUTCOMES:
Patient preference | 5 weeks
  Patient satisfaction, preference, and comfort with treatment

CONTACTS AND LOCATIONS:
Locations (1):
- McCabe Vision Center, Murfreesboro, Tennessee, United States